CLINICAL TRIAL: NCT01003431
Title: A Randomized, Open-Label Clinical Study to Assess the Immunogenicity and Safety of Whole-Cell Pertussis Containing Vaccine When Administered Concomitantly With RotaTeq™ or Rotarix™ in Healthy Infants in South Africa
Brief Title: A Study of the Immunogenicity and Safety of Whole-Cell Pertussis Containing Vaccine Administered Concomitantly With RotaTeq™ (V260) or Rotarix™ (V260-036)(WITHDRAWN)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V260-036; V260-036
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Rotavirus Gastroenteritis; Diphtheria; Tetanus; Pertussis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Rotavirus Vaccines; Diphtheria-Tetanus-acellular Pertussis Vaccines

ARMS (3):
- 1 (Experimental): RotaTeq™ + DTwP
  Interventions: Biological: Rotavirus Vaccine, Live, Oral, Pentavalent
- 2 (Active Comparator): Rotarix™ + DTwP
  Interventions: Biological: Comparator: Rotarix™ administered concomitantly with Tritanrix™ HepB (DTwP)
- 3 (Active Comparator): RotaTeq™ + DTaP
  Interventions: Biological: Comparator: RotaTeq™ administered concomitantly with INFANRIX™ (DTaP)

INTERVENTIONS:
Biological: Rotavirus Vaccine, Live, Oral, Pentavalent — [Intervention name: RotaTeq™ administered concomitantly with Tritanrix™ HepB (DTwP)] Three 2.0 mL oral doses of RotaTeq™ and three 0.5 mL intramuscular injections of Tritanrix™ HepB will be given at the same time with about 1 month between each administration.
  Arms: 1
Biological: Comparator: Rotarix™ administered concomitantly with Tritanrix™ HepB (DTwP) — Two 1.0 mL oral doses of Rotarix™ and three 0.5 mL intramuscular injections of Tritanrix™ HepB will be given at the same time with about 1 month between each administration (the second administration will be Tritanrix™ HepB only).
  Arms: 2
Biological: Comparator: RotaTeq™ administered concomitantly with INFANRIX™ (DTaP) — Three 2.0 mL oral doses of RotaTeq™ and three 0.5 mL intramuscular injections of INFANRIX™ will be given at the same time with about 1 month between each administration.
  Arms: 3

SUMMARY:
This study will evaluate the immunogenicity and safety of the pertussis component of DTwP (whole-cell pertussis containing vaccine) when administered concomitantly with RotaTeq™ or Rotatrix™.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants

Exclusion Criteria:

* History of abdominal disorders, intestinal folding, or abdominal surgery
* Impaired immune system
* Prior administration of any rotavirus vaccine or DTwP/DTaP
* Fever of >= 38.1C (100.5F) at the time of vaccination
* History of prior rotavirus infection, chronic diarrhea, or failure to thrive
* Evidence of active gastrointestinal illness

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2010-08 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) for Pertussis Toxoid | 1 month post dose 3

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) for rotavirus serotypes G1, G2, G3, G4 and P1A | 1 month post dose 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC